CLINICAL TRIAL: NCT06401460
Title: Gansu University of Chinese Medicine
Brief Title: Yannianjiuzhuan Method and Reverse Breathing Training to Improve Constipation in Elderly Patients With Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junfang Miao (Other)
Responsible Party: Sponsor-Investigator, Junfang Miao, Principal Investigator, Gansu University of Chinese Medicine
Organization: Gansu University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1774164090@qq.com
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Constipation; Coronary Heart Disease
MeSH Terms: conditions — Constipation; Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Yannianjiuzhuan method combined with reverse breathing training.
  Interventions: Other: Yannianjiuzhuan method combined with reverse breathing training
- Control group (Experimental): The control group received standard care in accordance with the "Constipation Nursing Protocol for Cardiology Patients," which included basic care, disease education, dietary and exercise guidance, bowel movement and psychological counseling .
  Interventions: Other: Yannianjiuzhuan method combined with reverse breathing training

INTERVENTIONS:
Other: Yannianjiuzhuan method combined with reverse breathing training — Timing of Operations
  1. Reverse Abdominal Breathing: Performed from 9:00 AM to 11:00 AM and from 7:00 PM to 9:00 PM daily, one inhalation and one exhalation constituting one cycle, with 30 cycles per training session, twice a day, over a period of ten days.
  2. Yannian Jiuzhuan Method: Conducted daily from 7:00 AM to 9:00 AM and from 9:00 PM to 11:00 PM, twice a day, for a duration of ten days.

SUMMARY:
Primary Purpose:

The primary purpose of this study is to evaluate the effectiveness of the Yannianjiuzhuan method combined with reverse abdominal breathing in improving symptoms of constipation, anxiety, sleep quality, and overall quality of life in elderly patients with coronary heart disease and constipation.

Study Phase:

As this research involves a non-pharmacological intervention, it is categorized as Not Applicable (N/A).

Intervention Model:

Parallel Assignment. Patients are divided into two groups; one receives standard care, while the other receives standard care supplemented by the Yannianjiuzhuan method combined with reverse abdominal breathing.

Number of Arms:

Two arms are involved in the study. One arm serves as the control group receiving standard care, and the other as the experimental group receiving standard care plus the Yannianjiuzhuan method combined with reverse abdominal breathing.

Masking:

This study employed a double-blind (assessors and statisticians), randomized, parallel-controlled trial design to enhance the credibility of the results and to minimize bias.

Allocation:

Using simple random sampling, small folded papers marked with the numbers "1" and "2" were placed in an opaque box. Each patient drew a paper in sequence of enrollment; those drawing a "1" were assigned to the control group, and those drawing a "2" to the experimental group, with each group comprising 35 participants.

Enrollment:

A total of 70 patients were initially recruited, with 67 completing the study. The control group had one participant drop out due to early hospital discharge related to the pandemic, affecting data collection completeness. In the experimental group, one participant was excluded due to undergoing colonoscopy and taking related laxative medications during the treatment, and another due to early hospital discharge caused by the pandemic. Thus, data from three participants were excluded from the final analysis due to insufficient treatment duration (less than two-thirds of the planned intervention), resulting in 34 participants in the control group and 33 in the experimental group being analyzed, equating to a dropout rate of approximately 4.3%, which is within acceptable statistical limits.

Study Classification:

This study focuses on efficacy assessment. It particularly evaluates the effectiveness of the Yannianjiuzhuan method combined with reverse abdominal breathing in alleviating symptoms of constipation, anxiety, improving sleep quality, and enhancing the quality of life among elderly patients with coronary heart disease and constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for chronic stable coronary heart disease and constipation .
2. Aged 60 years and above but below 80 years.
3. Heart function classified as ≤ Class 2.
4. Clear consciousness, no language barriers, free of dementia or psychiatric history, and willing to comply with treatment.
5. Voluntarily participating in the study and has signed the informed consent form.

Exclusion Criteria:

1. Patients participating in other trials that could affect the results of this study.
2. Patients with organic constipation, refractory constipation, or fecal incontinence.
3. Patients with significant physical mobility impairments.
4. Patients suffering from severe metabolic diseases, cardiopulmonary diseases, hematological diseases, or psychiatric disorders.
5. Patients who have undergone abdominal surgery or other conditions unsuitable for abdominal massage within the past six months.
6. Patients who have taken medications affecting digestive functions and bowel movement in the past week.
7. Patients who underwent lumbar surgery within the past six months.
8. Patients assessed by doctors as having severe constipation symptoms, which could potentially worsen their condition.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
PAC-SYM | Before the intervention，after 3 days of intervention，and after 10 days of intervention.
  Patient Assessment of Constipation Symptoms (PAC-SYM) : This scale assesses the clinical presentation and severity of constipation across three dimensions: abdominal, rectal, and stool symptoms, with a total of 12 items. Using a Likert 5-point scoring system, higher scores indicate more severe symptoms.
Bristol Stool Scale | Before the intervention，after 3 days of intervention，and after 10 days of intervention.
  Bristol Stool Scale: This scale is used to evaluate the characteristics of stool, with seven types ranked; lower scores denote harder stools, indicating more severe constipation.
SAS | Before the intervention and after 10 days of intervention.
  Self-Rating Anxiety Scale (SAS) : This scale is applicable to a broad population and assesses 20 items including anxiety and fear, using a Likert 4-point scoring system. Higher scores reflect greater anxiety levels.
PSQI | Before the intervention and after 10 days of intervention.
  Pittsburgh Sleep Quality Index (PSQI) : This index evaluates patient sleep quality across 24 items spanning seven dimensions. Higher scores indicate more severe sleep quality issues.
PAC-QoL | Before the intervention and after 10 days of intervention.
  Patient Assessment of Constipation Quality of Life (PAC-QoL) : Encompassing 28 items, this scale covers the dimensions of worry/concern, physical discomfort, psychosocial impacts, and satisfaction. Higher scores suggest greater impact on patients' quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Chengguanqu, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Undecided